CLINICAL TRIAL: NCT04947540
Title: Hematological and Biochemical Markers of Iron Status in Thalassemic Children Receiving Multiple Blood Transfusion
Brief Title: Iron Status in BTM With Blood Transfusion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Mohamed Rashed Gad, principle investigator, Assiut University
Other Study IDs: IS in BTM patients
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the possible role of iron overload as a cause of liver dysfunction in thalassemic childrens receiving multiple blood transfusion and its correlation with serum aminotransferases.

DETAILED DESCRIPTION:
Thalassemia is derived from the Greek words, thals, which means sea, and emia, which means blood, signifying that it is more common in the Mediterranean region . Globally, among humans, thalassemia is the commonest single-gene disorder. It is defined as a group of inherited disorders characterized by decreased or absent beta globin chain synthesis, leading to a reduced level of hemoglobulin (Hb) in the red blood cells . Specifically in developing countries, thalassemia is a huge health dilemma.

-Beta Thalassemia is the most common chronic hemolytic anemia in Egypt (85.1%) with an estimated carrier rate of 9-10.2%.

Blood transfusion is the primary way of treating thalassemia; it allows the normal growth of the child as well as restrains abnormal erythropoiesis . Iron-chelating agents should be used properly;otherwise, multiple blood transfusions can lead to iron overload. Yet, with no blood transfusion, the increase rate of erythropoiesis intensifies dietary iron absorption from the gut, leading to a severe form of iron overload .

iron overload can result in serious damage to various organs, for example, by depositing in the liver, heart, and various other endocrine glands along with endocrine organ failure. .

During the last years, liver disease has emerged as a major cause of mortality in patients with B- thalassemia major (TM).

The liver is the only site for ferritin and transferrin synthesis, as well as the primary organ for iron storage.

The liver has the maximum capacity to store excess iron in the body, and various other organs, as well as the liver, are very susceptible to damage as a result of iron toxicity.

The correlation between serum ferritin and hepatic iron concentration has been reported in multiple blood-transfused thalassemia patients .

Thalassemia major patients who undergo routine transfusion have an increased risk of acquiring transfusion-transmitted infections (TTI), including hepatitis B and C. These diseases have serious implications and may affect the serum ferritin and aminotransferase levels of thalassemia major patients.

Although the risk of post-transfusion hepatitis C virus (HCV) infection dropped significantly after the national screening of blood in 1993, more than 20% of children who were multitransfused after that date were HCV-RNA positive .

In Egypt, prevalence rate of HCV antibodies seropositivity in thalassemic children at 2011was 51.7% while in the study of El-Faramawy (2012) , a prevalence of 48 % was reported.

Iron overload and hepatitis-C virus (HCV) infection, have been implicated in the evolution of liver disease, in patients with transfusion-dependent beta-thalassaemia major (BTM). The impact of these factors and liver with BTM, has not been extensively studied yet.

Hepatitis virus C infection is the main risk factor for liver injury in transfusion-dependent thalassemics . Dimitrios (2013) on the other hand suggested that in the late stages of liver disease in BTM patients, iron overload may be the critical determinant, since fibrosis is related to the minimal haemosiderosis, independently of HCV history. Injury to the liver, whether acute or chronic, eventually results in an increase in serum concentrations of Alanine transaminase (ALT) and Aspartate transaminase (AST)

ELIGIBILITY:
Inclusion Criteria:

* Thalassemic patients of both sex.
* Beta-thalassemia major patients diagnosed Clinical and laboratory .
* Age 5 : 18 years.
* Undergoing multiple blood transfusion.

Exclusion Criteria:

* -Age less than 5 years.
* Acute illness as fever and infections.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: all cases diagnosed as thalassemia major attending to thalassemic center at hematological department at Assuit university childern hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Hematological and biochemical markers of Iron status in thalassemic children receiving multiple blood transfusion | baseline
  Assessment the possible role of iron overload as a cause of liver dysfunction in thalassemic childrens receiving multiple blood transfusion and its correlation with serum aminotransferases.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Ghazally, professor, Study Director — Egypt

REFERENCES:
- [Background] Al-Moshary M, Imtiaz N, Al-Mussaed E, Khan A, Ahmad S, Albqami S. Clinical and Biochemical Assessment of Liver Function Test and Its Correlation with Serum Ferritin Levels in Transfusion-dependent Thalassemia Patients. Cureus. 2020 Apr 7;12(4):e7574. doi: 10.7759/cureus.7574. PMID 32391223
- [Background] Amjad F, Fatima T, Fayyaz T, Khan MA, Qadeer MI. Novel genetic therapeutic approaches for modulating the severity of beta-thalassemia (Review). Biomed Rep. 2020 Nov;13(5):48. doi: 10.3892/br.2020.1355. Epub 2020 Sep 2. PMID 32953110
- [Background] Salama KM, Ibrahim OM, Kaddah AM, Boseila S, Ismail LA, Hamid MM. Liver Enzymes in Children with beta-Thalassemia Major: Correlation with Iron Overload and Viral Hepatitis. Open Access Maced J Med Sci. 2015 Jun 15;3(2):287-92. doi: 10.3889/oamjms.2015.059. Epub 2015 May 28. PMID 27275237